CLINICAL TRIAL: NCT01929421
Title: A Phase II Trial of Salvage Treatment With Gemcitabine and S-1 Combination in Patients With Heavily Treated Advanced Colorectal Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Hee Kyung Ahn, Assistant Professor, Gachon University Gil Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-GIRBA-2075
Record Dates: First submitted 2013-08-19; First posted 2013-08-28 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Advanced Colorectal Cancer
Keywords: colorectal cancer; gemcitabine; S-1
MeSH Terms: conditions — Colorectal Neoplasms

ARMS (1):
- Gemcitabine/ s-1 (Experimental)
  Interventions: Drug: Gemcitabine/S-1

INTERVENTIONS:
Drug: Gemcitabine/S-1

SUMMARY:
To assess the efficacy and safety of salvage tratment with Gemcitabine and S-1 Combination in metastatic colorectal cancer

ELIGIBILITY:
Inclusion Criteria:

* non resectable colorectal adenocarcinoma.
* disease progression during or within 6months after treatment with irinotecan and oxaliplatin contaning regimens.
* estimated life expectancy of more than 3 months.
* ECOG status 2 or lower

Exclusion Criteria:

* other tumor type than adenoarcinoma.
* presence or history of CNS metastasis.
* evidence of gastrointestinal bleeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-12; Primary Completion 2013-06 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Response rate | 1year

SECONDARY OUTCOMES:
overall survival | 1year
number of participants with adverse events | 1year

CONTACTS AND LOCATIONS:
Locations (1):
- Gachon University Gil Medical Center, Incheon, South Korea